CLINICAL TRIAL: NCT00449813
Title: The CONQUEST-Study. Evaluation of Clinical Endpoints for Treatment-induced Changes in GERD-related Symptoms
Brief Title: The CONQUEST-Study. Evaluation of Clinical Endpoints for Treatment-induced Changes in GERD-related Symptoms (BY1023/NL511)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inclusion-rate does not seem feasible anymore to obtain te required number of patients before the end of the trial.
Sponsor: Takeda (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/NL511
Record Dates: First submitted 2007-03-02; First posted 2007-03-21 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Gastroesophageal Reflux Disease; Non-erosive Reflux Disease
Keywords: Gastroesophageal reflux disease (GERD); Non erosive reflux disease (NERD)
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. (Active Comparator): 40 mg Pantoprazole
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — 40 mg Pantoprazole

SUMMARY:
The aim of the study is to compare two different endpoint measures: heartburn as assessed by the physicians versus gastroesophageal reflux disease (GERD)-related symptoms as assessed by the patient using the ReQuest™ questionnaire. The assessment is made in GERD-patients treated with a daily dose of 40 mg oral pantoprazole over an 8-week period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Outpatients of at least 18 years of age
* History of GERD-related symptoms of at least 6 months prior to baseline visit
* Endoscopically-confirmed GERD or non-erosive GERD

Exclusion Criteria:

* Zollinger-Ellison syndrome or other gastric hypersecretory condition
* Acute peptic ulcer and/or ulcer complications
* Pyloric stenosis
* Severe or unstable cardiovascular, pulmonary, and/or endocrine disease
* Pregnancy, breast feeding, intention to become pregnant during the course of the study or lack of reliable contraception in women of child-bearing potential
* Intake of any medication for the purpose of eradication of Helicobacter pylori (H. pylori) within the last 28 days prior to study start
* Intake of systemic glucocorticoids or non-steroidal anti-inflammatory drugs including cyclooxygenase-2 (COX-2) inhibitors for more than 3 consecutive days within the last 28 days prior to study start; with the exception of acetylsalicylic acid not more than 150 mg per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Rate of misclassification on day 14 based on heartburn as assessed by the investigator compared to symptom assessment by the patient using the ReQuest™-gastrointestinal (GI) questionnaire | 8 weeks

SECONDARY OUTCOMES:
Rate of misclassification on day 14 based on acid regurgitation as assessed by the investigator compared to symptom assessment by the patient using the ReQuest™-GI questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: M. Oudkerk Pool, Prof., Principal Investigator — Isala Klieniken, Zwolle, The Netherlands
Locations (13):
- Netherlands (3):
  - Altana Pharma/Nycomed, BT Oss
  - Altana Pharma/Nycomed, Den Helder
  - Altana Pharma/Nycomed, EH Geldrop
- Switzerland (10):
  - Altana Pharma/Nycomed, Basel
  - Altana Pharma/Nycomed, Biel/Bienne
  - Altana Pharma/Nycomed, Bülach
  - Altana Pharma/Nycomed, Locarno, TI.
  - Altana Pharma/Nycomed, Lucerne
  - Altana Pharma/Nycomed, Reinach
  - Altana Pharma/Nycomed, Sion
  - Altana Pharma/Nycomed, Thun
  - Altana Pharma/Nycomed, Winterthur
  - Altana Pharma/Nycomed, Zurich